CLINICAL TRIAL: NCT01868971
Title: EndoRings™ - Clinical Protocol
Brief Title: Clinical Study to Establish the Feasibility and Usability of the EndoRings™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EndoAid (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CSDPR100
Record Dates: First submitted 2013-05-29; First posted 2013-06-05 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Colon Cancer; Bowel Cancer; Colorectal Cancer
Keywords: EndoRings
MeSH Terms: conditions — Colonic Neoplasms; Intestinal Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Colonoscopy procedure with the EndoRings (Other): Colonoscopy procedure using an add-on device (EndoRings) that is attached to the distal tip of the endoscope
  Interventions: Device: EndoRings

INTERVENTIONS:
Device: EndoRings — Colonoscopy procedure, standard endo-therapy interventions will be performed in accordance with physician's evaluation

SUMMARY:
The purpose of this prospective clinical study is to establish the feasibility and usability of the ENDORINGS™ when used during standard colonoscopy procedure.

DETAILED DESCRIPTION:
The EndoAid Ltd. EndoRings is used during endoscopy procedures. The EndoRings is a short silicon rubber tube with flexible circular wings that attaches to the distal end of the endoscope to facilitate endoscopic therapy.

The EndoRings is designed to fit specific endoscopes (as designated on the packaging), and is supplied sterile following ETO sterilization and is single use only.

Indications for Use:

To be attached to the distal end of the endoscope to facilitate endoscopic therapy, to be used for the following:

* Keeping the suitable depth of endoscope's view field
* Helping the endoscope with being inserted into the gastrointestinal tract

Patient Population: The study population is comprised of patients indicated for colonoscopy.

Study Design: Single-center study. A single treatment group of 60 patients. No. of Patients: Up to sixty (60) treated patients will be enrolled in the study.

Primary Endpoints:The primary endpoint is reaching the cecum of the colon with the ENDORINGS™.

Secondary Endpoints / Other Outcomes:

1. Incidence of complications (number of complications)
2. Ability to complete s therapeutic interventions as biopsies, polypectomies, APC etc.
3. Procedure time.
4. Ease of scope insertion, advancement and withdrawal.
5. Ability to center the scope inside the gastrointestinal tract.
6. Subjective evaluation of the additional area screened by the physician (recorded in the source documents by a questionnaire).
7. Patient satisfactory (by a follow up phone-call in which questionnaire with VAS scale will be filled out).

ELIGIBILITY:
Inclusion Criteria:

Any subject who meets all of the following criteria may be included in this study:

* Subject between the ages of 18 and 70
* The patient is undergoing colonoscopy for screening, or for surveillance in follow-up of previous polypectomy or for diagnostic workup;
* Written informed consent must be available before enrollment in the trial
* For women with childbearing potential, adequate contraception

Exclusion Criteria:

Any subject who meets any of the following criteria will not be included in this study:

* Patients with a history of colonic resection;
* Patients with inflammatory bowel disease;
* Patients with a personal history of polyposis syndrome;
* Patients with suspected chronic stricture potentially precluding complete colonoscopy;
* Patients with diverticulitis or toxic megacolon;
* Patients with a history of radiation therapy to abdomen or pelvis;
* Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is reaching the cecum of the colon with the ENDORINGS™. | 24 hours post procedure

SECONDARY OUTCOMES:
1. Incidence of complications (number of complications) | 24 hours post procedure
  Known complications include:
  * Perforation;
  * Severe abdominal pain;
  * Infection;
  * Bleeding (other than expected minor bleeding due to therapeutic procedures e.g. polypectomy);
  * Inducing inflammation of diverticulum
  * Arrhythmia, bradycardia, hypotension, hypoxia
  * Death A complication is defined as any one of the above complications as well as any other unexpected complication requiring medical intervention beyond that of the standard procedure. All adverse events will be reported and treated as per the standard clinical practices.
  A telephone call should be made to the patient at 24 hour post- procedure, to assess post-examination adverse events.
2. Ability to complete s therapeutic interventions as biopsies, polypectomies, APC etc. | 24 hours post procedure
  Whenever a polyp or other abnormality is detected, the endoscopist will perform biopsy, polypectomy or other evaluation or therapy as appropriate. The clinical investigator will use his/her clinical judgment on the safety of polyp removal/biopsy.
3. Procedure time. | During procedure
  Procedural times for each colonoscopy procedure:
  1. Time for intubation to the cecum
  2. Time for withdrawal from the cecum to the anal verge
  3. Total procedure time
4. Ease of scope insertion, advancement and withdrawal. | During procedure
  Physician's subjective evaluation will be recorded in the source documents by a questionnaire.
5. Ability to center the scope inside the gastrointestinal tract. | During procedure
  Physician's subjective evaluation will be recorded in the source documents by a questionnaire.
6. Subjective evaluation of the additional area screened by the physician. | During procedure
  Physician's subjective evaluation will be recorded in the source documents by a questionnaire.
7. Patient satisfactory. | During procedure
  A telephone call should be made to the patient at 24 hour post- procedure, to assess patient satisfactory by completing a VAS scale questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Gralnek, Prof., Principal Investigator — Attending Physician at Elisha Hospital, Haifa, Israel ~~~~~ Chief, Hospital-Wide Ambulatory Care Services Head, GI Outcomes Unit and Senior Physician Department of Gastroenterology Rambam Health Care Campus Rappaport Faculty of Medicine, Technion-Israel
Locations (1):
- Elisha Medical Center, Haifa, Please Select, Israel